CLINICAL TRIAL: NCT05483556
Title: Brain Network Plasticity in Aphasic Patients Associated With Combined Speech Therapy and Transcranial Direct Current Stimulation
Brief Title: tDCS Effects on Brain Plasticity in Aphasia Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Min Wong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20220211001
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Aphasia; Stroke
Keywords: tDCS; MRI; Aphasia; Stroke; Speech therapy
MeSH Terms: conditions — Aphasia; Stroke; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant, outcome accessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): Five post-stroke patients will be allocated by the flip the coin method to the experimental group. Participants will receive anodal tDCS stimulation for 20 minutes
  Interventions: Device: Real tDCS
- Sham tDCS (Sham Comparator): Five participants will be allocated by the flip coin method to the sham comparator group. Participants will receive the tDCS stimulation for the 30s
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Real tDCS — An anodal high-definition tDCS of 2 mA lasting for 20 minutes will be delivered to the left inferior frontal gyrus during speech therapy.
  Arms: Real tDCS
Device: Sham tDCS — An anodal high-definition tDCS of 2 mA lasting for 30 seconds will be delivered to the left inferior frontal gyrus during speech therapy.
  Arms: Sham tDCS

SUMMARY:
The efficacy of conventional speech therapy alone for aphasia recovery is inconclusive. The prospective study will monitor the effects of combined language therapy and tDCS through structural and functional MRI.

DETAILED DESCRIPTION:
The efficacy of conventional speech therapy alone for aphasia recovery is inconclusive. The prospective study will monitor the effects of combined language therapy and tDCS through structural and functional MRI.

This randomized, placebo-controlled, double-blinded pilot study will recruit ten chronic stroke patients with Broca's Aphasia randomly assigned either to sham or an anodal tDCS groups. Following speech and language assessment, all the participants will receive 20 minutes of individualized language therapy daily for ten days in two consecutive weeks. Simultaneously, the treatment group will receive 20 minutes of 2mA anodal HD-tDCS over the left IFG, while the sham group will receive the 30s of 2mA anodal HD-tDCS. Structural, resting state and task activated functional MRI will be performed. Data acquisition will be performed before, immediately after and two months after the treatment.

Repeated measure ANOVA for changes in picture-naming accuracy and response time will be performed as a within-subject factor between sham and anodal tDCS. Pearson's correlation coefficient of left IFG and its homolog in the right hemisphere through Independent component analysis (ICA) of low-frequency fluctuations in resting-state and task activated state will be compared for functional connectivity analysis for IFG and other major languages hubs for oral language production between groups.

ELIGIBILITY:
Inclusion Criteria:

1. History of a single unilateral left-hemispheric stroke,
2. Right handedness
3. Demonstrated features of Broca's Aphasia
4. Cantonese speaker
5. Comprehension sufficient to carry out tasks
6. No history of other neurological diseases

Exclusion Criteria:

1. Aphasia due to reasons other than Stroke, Traumatic brain injury
2. Bilateral or multiple brain lesions
3. Wernicke's aphasia and other speech disorders, degenerative, psychiatric or metabolic disorders
4. Deaf, blind, pregnant/ or preparing for pregnancy, cognitive issues, tattoos
5. Have cochlear implants, pacemaker, surgical nails for bone fracture, artificial joints, dental braces, dentures
6. Taking anti-depressant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Picture naming | Change before, immediately after and two months after the treatment
  Picture-naming accuracy and response time for each stimuli will be determined perceptual and calculated using praat software

SECONDARY OUTCOMES:
Imaging analysis | Change before, immediately after and two months after the treatment.
  Mapping changes in functional connections of language networks, inter-hemispheric and intra-hemispheric regions of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Min Ney Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong